CLINICAL TRIAL: NCT02934919
Title: Evaluation of Nalmefene in Impulse Control Disorders in Parkinson's Disease: A Prospective Open Label Study
Acronym: Nalmefene TCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0286; 2016-002805-21 (Other: 2016-002805-21)
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Impulse Control Disorders; Parkinson Disease
Keywords: Nalmefene; Impulse control disorders; Parkinson's disease; Tolerance; Efficacy
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Parkinson Disease | interventions — nalmefene

ARMS (1):
- nalmefene (Experimental)
  Interventions: Drug: Nalmefene

INTERVENTIONS:
Drug: Nalmefene — 30 patients with ICDs, will be treated with 18 mg per day of nalmefene during 3 months

SUMMARY:
Impulse control disorders (ICDs) (such as pathological gambling, hypersexuality, compulsive shopping …) are an increasingly recognized psychiatric complications in Parkinson's disease (PD). Therapeutic management of these disorders is important since they have an impact on patient quality of life. Dopamine agonists play a key role in the emergence of ICD.

Animal models and imaging underline the implication of opioid system in the genesis of ICD.

An opioid antagonist, the naltrexone, has been studied to treat ICDs in PD. Papay and al 2014 have found that patients treated by naltrexone showed an interesting decrease of their ICDs measured by the QUIP RScale. Nevertheless, naltrexone has shown adverse effects such as increasing hepatic liver enzymes. Nalmefene has no known hepatic adverse effects. Nalmefene is an opioid antagonist that has an antagonist action on μ and δ receptors, but also an agonist action on κ receptor. Grant and al 2006 has shown significant reduction of the severity of pathological gambling in patients treated with nalmefene.

The primary purpose is to evaluate the efficacy and the safety of nalmefene in the treatment of ICDs in PD.

DETAILED DESCRIPTION:
In this open study, 30 patients with ICDs, will be treated with 18 mg per day of nalmefene during 3 months.

Patients will be evaluated 2 times: at inclusion visit (J0) and 3 months after (at the end of the study, +3months).

At each time, patients will have :

* a clinical and neurological evaluation
* neuropsychological tests for cognitive, depression and TCI evaluations.
* blood sample to test hepatic and renal functions
* tolerance evaluation with a list of adverse events/effects

Patients will be contacted 3 times by phone: 2 weeks after inclusion, 1 month after inclusion and 2 months after inclusion, to note the presence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering of Parkinson's disease
* Male or Female aged from 18 to 80 years old
* Diagnosis of ICDs with the Ardouin Scale of Behavior in Parkinson's Disease (ASBPD) with a score of at least 2 on one of the Item of hyperdopaminergic symptoms
* No modification of the treatments for PD since 3 months
* No modification of parameters of deep brain stimulation since 6 months
* Patients who understood and signed the consent form
* Patients having a social security

Exclusion Criteria:

* Contraindication to nalmefene (Patients receiving opioid antalgics, antecedent of opioid dependence, dopamine agonist withdrawal syndrome, opioid consumption, patient receiving methadone or buprenorphine, severe hepatic failure, severe renal failure, antecedent of alcohol withdrawal, galactose intolerance, lactose deficit or glucose malabsorption, pregnant women)
* Cognitive impairment with Mini Mental Score < 26
* Psychiatric comorbidities (bipolar disease, schizophrenia)
* Patient participating in another therapeutic study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Tolerance of Nalmefene measured by the dropout rate secondary to adverse effects | at + 3months
Efficacy of Nalmefene measured by the change from baseline of the QUIP-RS | at + 3months

SECONDARY OUTCOMES:
Change from baseline of the cognitive state assessed by the Montreal Cognitive Assessment scale | at +3 months
Change from baseline of the depression assessed by the Hamilton scale | at +3 months
Change from baseline of the motor severity assessed by the Unified Parkinson Disease Rating Scale at +3 months | at +3 months
Change from baseline of hepatic and renal function evaluated with blood samples at +3 months | at +3 months

CONTACTS AND LOCATIONS:
Overall Officials: Franck DURIF, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France